CLINICAL TRIAL: NCT06555198
Title: Promotion of Nurses' Lower Extremity Health by Foot(at)Work Intervention to Support Work Wellbeing
Brief Title: Promotion of Nurses' Lower Extremity Health by Foot(at)Work Intervention
Acronym: Foot(at)Work
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: The Hospital District of Satakunta (Other); Finnish Work Environment Fund (Other)
Responsible Party: Principal Investigator, Minna Stolt, professor (act.), PhD, University of Turku
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 230374
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-08

CONDITIONS: Lower Extremity Problem; Foot Deformities
MeSH Terms: conditions — Foot Deformities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Foot(at)Work intervention will be offered to participant sin the intervention group. The Foot(at)Work intervention lasts for 5 weeks. The intervention is constructed on electronic learning environment consisting of 5 themes illustrating self-care activities for common foot problems among nursing professionals. The idea of self-directed learning is to support nurses competence to self-care their lower extremities and thus, promote their work wellbeing in clinical nursing environments.
  Interventions: Behavioral: Foot(at)Work intervention
- Control group (No Intervention): The control group will work and live as usual.

INTERVENTIONS:
Behavioral: Foot(at)Work intervention — Foot(at)Work intervention is targeted for nurses working in clinical settings to promote their competence in lower extremity health self-care.
  Arms: Intervention group

SUMMARY:
The quasiexperimental study aims to analyse the effecs of Foot(at)Work intervention on nurses' lower extremity health. The Foot(at)Work intervention is in electronic format consisting of 5 themes. The idea is that the participants familiarizes with the foot health -related content. The primary outcome is knowledge about lower extremity self-care. Secondary outcomes are work well-being, lower extremity health and musculoskeletal health. The outcomes are measured before the intervention (M0), after the intervention (M1), one month after the intervention (M2), six months after the intervention (M3) and 12 months after the intervention (M4).

The purpose of the Foot(at)Work intervention is to support nurses ability to self-care their lower extremities. The intervention consists of text, videos, and pictures that educate nurses to self-care their lower extremities and to select proper footwear.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurse
* Working in the specialized health care in surgical or internal medicine wards of one certain hospital

Exclusion Criteria:

* Nursing students

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Knowledge of lower extremity self-care | before intervenion, right after the intervention, one, six and 12 months after the intervention
  Knowledge will be measured with self-administered questionnaira that contains 20 items (response options yes-no) about self-care for lower extremity problems.

SECONDARY OUTCOMES:
Self-assessed foot health | before intervenion, right after the intervention, one, six and 12 months after the intervention
  Self-Administered Foot Health Assessment Instrument (S-FHAI) will measure subjective self-assessment measure of current foot health with 22 items. Four subcategories were included: skin health (12 items), nail health (4 items), foot structure (5 items), and foot pain (1 item).
Musculoskeletal health | before intervenion, right after the intervention, one, six and 12 months after the intervention
  Nordic Musculoskeletal Questionnaire will be used as self-report measure to assess the impact of a musculoskeletal condition on an individual's functioning and on the impact of the condition on daily activities.
Self-perceived work ability | before intervenion, right after the intervention, one, six and 12 months after the intervention
  Work ability index: one question where respondent indicates the level of perceived current work ability. Range 1-10 where 1 indicates not capable of working - 10 best possible work ability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turku, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No